CLINICAL TRIAL: NCT03117972
Title: Chemotherapy Intensification in Patients With High Lactate Dehydrogenase Values and Soluble Syndecan-1 Levels
Brief Title: Chemotherapy Intensification in Patients With High Lactate Dehydrogenase Values and Soluble Syndecan1 Levels
Acronym: CLavSyn
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: enrollment too slow
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: API/2016/73
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; Biomarker; Chemotherapy intensification; Syndecan1; LDH; CD138
MeSH Terms: conditions — Colorectal Neoplasms | interventions — FOLFOXIRI protocol; Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil; Folfox protocol; IFL protocol; Bevacizumab; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A : FOLFOXIRI - bevacizumab (Experimental): FOLFOXIRI + bevacizumab, 12 cures following by maintenance chemotherapy (bevacizumab + LV5FU2 or bevacizumab-capecitabine) until disease progression or limiting toxicities
  Interventions: Drug: FOLFOXIRI; Drug: Bevacizumab; Drug: LV5FU2; Drug: Capecitabine
- Arm B: FOLFOX or FOLFIRI - bevacizumab (Active Comparator): FOLFOX or FOLFIRI + bevacizumab 12 cures following by maintenance chemotherapy (bevacizumab + LV5FU2 ou bevacizumab capecitabine) until disease progression or limiting toxicities
  Interventions: Drug: FOLFOX; Drug: FOLFIRI; Drug: Bevacizumab; Drug: LV5FU2; Drug: Capecitabine

INTERVENTIONS:
Drug: FOLFOXIRI — 12 cycles
  Other Names: Irinotecan; Oxaliplatin; Leucovorin; 5-Fluorouracil
  Arms: Arm A : FOLFOXIRI - bevacizumab
Drug: FOLFOX — 12 cycles
  Other Names: Oxaliplatin; 5-Fluorouracil
  Arms: Arm B: FOLFOX or FOLFIRI - bevacizumab
Drug: FOLFIRI — 12 cycles
  Other Names: Ironotecan; Leucovorin; 5-Fluorouracil
  Arms: Arm B: FOLFOX or FOLFIRI - bevacizumab
Drug: Bevacizumab — 12 cycles
Drug: LV5FU2 — Maintenance chemotherapy
Drug: Capecitabine — Maintenance chemotherapy

SUMMARY:
In first-line metastatic colorectal cancer (mCRC), baseline prognostic factors allowing death risk and strategy stratification are lacking. In this setting, a simple biological scoring system have recently been proposed, including LDH and CD138 binary status seric values, identifying one third of patients with worst prognostic.

Intensified-chemotherapy strategies, combining 5-fluorouracile, Oxaliplatin, Irinotecan and Bevacizumab, are beneficial for patients having a bad prognostic, defined by the BRAFV600E mutation, concerning 5-8% of first line mCRC.

For the 30% of patients with LDH-CD138 elevated score, the purpose of CLavSyn phase II study is to compare the PFS of one intensified arm (FOLFOXIRI Bevacizumab) to one standard chemotherapy arm, in order to better discriminate treatment strategies, at metastatic diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Performance status ECOG-WHO 0 or 1
* Histologically proved metastatic colorectal adenocarcinoma, with non-resectable metastases
* Adequate hematological, hepatic, and renal functions
* Signed written informed consent

Exclusion Criteria:

* Previous treatment (chemotherapy, targeted therapy, surgery) for metastatic disease
* History of autoimmune disease
* Acute infectious disease
* Known hypersensitivity grade 3-4 or contraindication to any of the study drugs
* Patient with any medical or psychiatric condition or disease which would make the patient inappropriate for entry into this study.
* Bevacizumab contraindication
* Brain metastases
* Other malignancy within the last 2 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer.
* Pregnancy, breast-feeding or absence of adequate contraception for fertile patients
* Patient under guardianship, curator or under the protection of justice.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | up to 4 years (3 years of inclusion and 12 months of follow up after the last patient included)
  Delay from the date of randomization to the disease progression (RECIST) or death from any cause whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Christophe BORG, Pr, Principal Investigator — Centre Hospitalier Universitaire de Besançon
Locations (10):
- France (10):
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Centre Hospitalier de Boulogne sur Mer, Boulogne-sur-Mer
  - CH de Colmar, Colmar
  - Institut de Cancérologie de Bourgogne, Dijon
  - CHRU de LILLE, Lille
  - Hôpital Nord Franche-Comté, Montbéliard
  - CHU de REIMS, Hôpital Robert Debré, Reims
  - Clinique Sainte Anne, Strasbourg
  - Centre Paul Strauss, Strasbourg
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jary M, Lecomte T, Bouche O, Kim S, Dobi E, Queiroz L, Ghiringhelli F, Etienne H, Leger J, Godet Y, Balland J, Lakkis Z, Adotevi O, Bonnetain F, Borg C, Vernerey D. Prognostic value of baseline seric Syndecan-1 in initially unresectable metastatic colorectal cancer patients: a simple biological score. Int J Cancer. 2016 Nov 15;139(10):2325-35. doi: 10.1002/ijc.30367. Epub 2016 Aug 13. PMID 27472156